CLINICAL TRIAL: NCT06597396
Title: A Phase 2a Randomized, Dose Ranging, Double-Blind, 3-Arm Study to Investigate Orally Administered Abrocitinib Compared With Placebo in Non-Hospitalized Symptomatic Adult Participants With Severe Fatigue From Post COVID Condition
Brief Title: Study to Investigate the Efficacy of Abrocitinib in Adult Participants With Severe Fatigue From Post COVID Condition/Long COVID
Acronym: CLEAR-LC
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Dan Barouch, Director of the Center for Virology and Vaccine Research, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2024P000700
Record Dates: First submitted 2024-09-12; First posted 2024-09-19 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Post-COVID Condition; Fatigue Symptom
Keywords: Long COVID; Post-COVID Condition; PCC; Fatigue
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Fatigue | interventions — abrocitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm 1: Abrocitinib 50 mg daily (Experimental): Participants will take 50 mg of abrocitinib daily for 12 weeks
  Interventions: Drug: Abrocitinib; Drug: Placebo
- Arm 2: Abrocitinib 100 mg once daily (Experimental): Participants will take 100mg of abrocitinib daily for 12 weeks
  Interventions: Drug: Abrocitinib
- Arm 3: Placebo (Placebo Comparator): Participants will take placebo daily for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Abrocitinib — 50 mg tablets
  Arms: Arm 1: Abrocitinib 50 mg daily; Arm 2: Abrocitinib 100 mg once daily
Drug: Placebo — Tablets
  Arms: Arm 1: Abrocitinib 50 mg daily; Arm 3: Placebo

SUMMARY:
The primary purpose of this phase 2a study is to compare the efficacy of abrocitinib to placebo in improving severe fatigue in non-hospitalized adults with symptomatic Post-COVID Condition (PCC) (also called Long COVID). We are also interested in learning if abrocitinib is effective in improving overall health status in people suffering from severe fatigue from PCC. Eligible participants with a confirmed history of COVID19 infection who also have PCC according to the World Health Organization definition, will be randomized to receive abrocitinib at a dose of 50 mg, 100 mg, or placebo by mouth daily for 12 weeks (84 days).

DETAILED DESCRIPTION:
Eligible volunteers will participate in six in-person visits at Beth Israel Deaconess Medical Center over 5 months. These visits include review of medical and medication history, answering questionnaires, blood, urine, and nasal swab specimen collection, physical exams, and contraceptive and medication counseling.

ELIGIBILITY:
Inclusion Criteria:

* History of confirmed COVID-19 infection
* PCC diagnosis according to the WHO definition as occurring in individuals with a history of probable or confirmed SARS CoV-2 infection, usually 3 months from the onset of COVID-19 that lasts for at least 2 months and cannot be explained by an alternative diagnosis
* Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures
* Capable of giving signed informed consent

Exclusion Criteria:

* Participants with acute and chronic infections, history of specific recurrent infections
* Suspected or confirmed active SARS-CoV-2 infection within past 30 days
* Some cardiac conditions
* Any current tobacco smoker or person who has smoked tobacco products within 12 months of screening, or former tobacco smoker ≥ 50 years old
* Known to be infected with Human Immunodeficiency Virus (HIV), Hepatitis B, or Hepatitis C, Herpes Virus, or Tuberculosis
* History of immunodeficiency
* Blood clotting conditions
* Must meet general screening laboratory criteria
* Allergy or other contraindication to any of the components of the study intervention
* Known prior participation in this trial or other trial involving abrocitinib
* Concurrent therapy with a JAK or TYK2 inhibitor
* Other protocol criteria apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2024-12-27 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in mean score for FACIT (Functional Assessment of Chronic Illness Therapy) Fatigue Scale | Baseline to Day 84
  To compare the efficacy of abrocitinib to placebo in improving severe fatigue in adults with symptomatic PCC

SECONDARY OUTCOMES:
Change from baseline for EQ(EuroQol)-5D-5L values and visual analog scale (VAS) score to Day 84 | Baseline to Day 84
  To compare efficacy of abrocitinib to placebo in improving health status in adults with symptomatic PCC
Change from baseline in PASC Symptom PRO (patient reported outcome) Instrument score to Day 84 | Baseline to Day 84
  To compare efficacy of abrocitinib to placebo in improving health status adults with symptomatic PCC
Safety-related clinical laboratory test abnormalities and related adverse events | Baseline to Day 84
  To describe the safety and tolerability of abrocitinib compared to placebo in the treatment of PCC in adults with symptomatic PCC
The difference in blood high sensitivity C-reactive protein (HSCRP) from baseline visit to Day 84 | Baseline to Day 84
  To compare the effect of abrocitinib to placebo for the treatment of symptomatic PCC in reducing HSCRP values

CONTACTS AND LOCATIONS:
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

REFERENCES:
- See also: Long COVID involves activation of proinflammatory and immune exhaustion pathways — https://www.nature.com/articles/s41590-025-02353-x